CLINICAL TRIAL: NCT02090075
Title: Apixaban Versus Warfarin in the Evaluation of Progression of Atherosclerotic Calcification and Vulnerable Plaque
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Matthew J. Budoff, Professor of Medicine, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21183-01
Record Dates: First submitted 2014-03-16; First posted 2014-03-18 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-03

CONDITIONS: Atrial Fibrillation
Keywords: cardiac Computed tomography; coronary calcification; intervention; warfarin; apixaban
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban; Warfarin

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- apixaban (Active Comparator): apixaban 5 mg or 2.5 mg po bid
  Interventions: Drug: apixaban
- warfarin (Placebo Comparator): warfarin with target INR of 2-3
  Interventions: Drug: warfarin

INTERVENTIONS:
Drug: apixaban — 5 po or 2.5 po bid.
  Other Names: eliquis
  Arms: apixaban
Drug: warfarin
  Other Names: Coumadin
  Arms: warfarin

SUMMARY:
Vitamin K-antagonists (VKA) such as warfarin are the most widely used blood thinners for irregular heart beats like atrial fibrillation. Several lines of evidence indicate, however, that these agents also cause calcification of vessels (hardening of the vessels). Vascular calcification is one of the recently revealed side-effects of warfarin therapy. We will be randomizing 66 patients to either take warfarin or a new blood thinner that works without affecting vitamin k (apixaban). Patients will undergo blood testing and a CT angiogram (non-invasive angiogram) at the beginning of the study, and then be followed for one year with quarterly visits including blood tests and given either warfarin or vitamin K. After one year, they will undergo another CT angiogram and examination and blood tests and the effect of apixaban and warfarin are tested to look at plaque and changes over time. Patients will be consented in a private room and the risks and benefits will be explained. The risks include the CT angiogram and the possibility of either remaining on warfarin therapy for another year (standard of care) or taking a medicine that doesn't require monitoring (apixaban) for one year. The CT angiograms will require some contrast and some radiation dose, which will be minimized as much as possible. A cardiologist will be present during each CT angiogram to minimize risk and ensure patient safety.

DETAILED DESCRIPTION:
The progression of atherosclerotic plaques characterized by various anatomic plaque composition changes has been acknowledged to be associated with increased plaque rupture, myocardial infarction and death. Coronary computed tomography angiography (CCTA) has emerged as a novel non-invasive modality with high diagnostic performance for detection and assessment of atheroma compared to invasive coronary angiography (ICA) and intravascular ultrasound (IVUS). Beyond stenosis severity, CCTA also permits anatomic quantification of numerous atheroscleroticStudy design This is a prospective, single-centered, randomized, open-label trial with blinded adjudication of results (plaque composition) designed to compare apixaban (2.5 mg or 5 mg BID per the current guideline) with warfarin (target international normalized ratio, 2.0 to 3.0) for 52 weeks on calcified plaque, coronary plaque composition and volume in patients with non-valvular AF.

Study population The targeted population included patients aged 18-84 years with non-valvular AF or flutter at enrollment or two more episodes of AF (as documented by electrocardiography) at least 2 weeks apart in the 12 months before enrollment. The inclusion and exclusion criteria were shown in detail in a recent paper. Subjects were enrolled from May 2014 to December 2015 and randomized into warfarin group (VKA_group) or apixaban group (Api_group). Of the 66 originally enrolled patients, 56 had complete data at final follow-up, including interpretable CCTA scans at baseline and follow-up. All subjects were followed up for a total 52 weeks.

Coronary CTA scan protocol All CT scans were performed with a 64-slice CT scanner (Lightspeed VCT; General Electric Healthcare Technologies, Milwaukee, WI, USA), or 256-slice CT scanner (Revolution CT; General Electric Healthcare Technologies, Milwaukee, WI, USA). Before CCTA, a prospective non-enhanced coronary calcium (CAC) scan was performed. For quantitative assessment of CAC, the Agatston score was calculated, using a 3 mm CT slice thickness and a detection threshold of ≥130 HU involving ≥1 mm2 area/lesion (3 pixels). CCTA was performed using a collimation of 64 × 0.625 mm or 256 × 0.625 mm and a rotation time of 0.4 s or 0.28 s. The tube current was 400-770 mA (depending on body weight), at 100-120 kV. Contrast material at a flow rate of 5.0 mL/s was administered in the antecubital vein, with volumes depending on the total scan time (60-80 mL). In the absence of contraindications, patients with a heart rate ≥60 bpm were administered 50-100 mg metoprolol oral and up to 40 mg metoprolol intravenous if needed. Interpretation was performed by expert reading by an experienced cardiologist (M.J.B) blinded to all clinical data.

plaque phenotypes, plaque burden and ability to differentiate between various plaque types. Also, recent technology providing low radiation dose for CCTA with approximately < 1-3mSv allows us to investigate the effects of different therapies using serial CCTA.

Warfarin, a vitamin K antagonist (VKA) and one of the most commonly used oral anti-coagulants, has been showed to increase vascular calcification leading to increased cardiovascular (CV) events. However, apixaban, a direct Factor Xa inhibitor, has no interaction with vitamin K and its effect on the progression of atherosclerotic plaques is still unknown. The potential benefit of avoiding VKA therapy and the favorable effects of factor Xa inhibitors may contribute to a reduction in CV events. We aimed to compare apixaban with warfarin on progression of coronary plaque composition and volume in non-valvular AF patients using CCTA.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients with atrial fibrillation or flutter
* Age 18-84 years
* Willingness to participate in the study and ability to sign informed consent.

Exclusion Criteria:

* Atrial fibrillation due to a reversible cause
* moderate or severe mitral stenosis
* conditions other than atrial fibrillation that require anticoagulation (e.g., a prosthetic heart valve)
* A need for aspirin at a dose of >165 mg a day or for both aspirin and P2Y-inhibitor
* Serious bleeding event in the previous 6 months or a high risk of bleeding (eg, active peptic ulcer disease)
* a platelet count of <100,000/mm3 or hemoglobin level of <10 g/dL
* stroke within the previous 10 days
* documented hemorrhagic tendencies, or blood dyscrasias
* Renal insufficiency (serum creatinine level of 12.5 mg per deciliter or calculated creatinine clearance of <50 ml per minute)
* Weight in excess of 325 pounds
* Resting hypotension (systolic blood pressure of <90mmHg) or resting hypertension (systolic blood pressure of >170mmHg or diastolic blood pressure of >110 mmHg)
* History of active malignancy requiring concurrent chemotherapy
* Known allergy to iodinated contrast material
* pregnancy, women of childbearing potential unwilling to use adequate contraception.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2014-09; Primary Completion 2016-12-27 (Actual); Study Completion 2017-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Budoff, MD, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (1):
- Los Angeles Biomedical Research Institute, Torrance, California, United States

REFERENCES:
- [Derived] Win TT, Nakanishi R, Osawa K, Li D, Susaria SS, Jayawardena E, Hamal S, Kim M, Broersen A, Kitslaar PH, Dailing C, Budoff MJ. Apixaban versus warfarin in evaluation of progression of atherosclerotic and calcified plaques (prospective randomized trial). Am Heart J. 2019 Jun;212:129-133. doi: 10.1016/j.ahj.2019.02.014. Epub 2019 Mar 13. PMID 31002997

RESULTS

PARTICIPANT FLOW:
Groups:
- Warfarin: warfarin with target INR of 2-3
  warfarin
Period: Overall Study
Arm/Group | Apixaban | Warfarin
Started | 33 | 33
Completed | 26 | 30
Not Completed | 7 | 3

BASELINE CHARACTERISTICS:
Population: all patients who were initially enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Warfarin | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 33 | 66
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (2.4) | 60 (1.9) | 57 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 19 | 23 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 5 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 13 | 23
  White | 20 | 15 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 33 | 66
coronary calcium [Number; unit: participants with coronary calcium] | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Coronary Artery Calcium (CAC) Score
Description: amount of calcification measured by Agatston Score. The range of values for the Agatston score is 0-10000. Higher score is worse outcome.
Time Frame: 1 year
Population: all with follow up scans
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 26 | 30
units on a scale | 66 (129.9) | 31 (61.5)

2. Secondary Outcome: Coronary Plaque on CT Angiography
Description: To evaluate if treatment with apixaban therapy, as compared to warfarin therapy, will modify the progression, regression and stabilization of coronary atherosclerosis. Modifications will include differences in plaque volume, composition and arterial remodeling; as well as new atherosclerosis formation. The scale is based upon volume of plaque in the coronary arteries, with zero being no plaque and a higher number being more plaque. There is no scale or maximum measure, this is a linear measure of atherosclerosis volume in the coronary arteries and more is worse. None is best, any plaque is considered worse, and a higher plaque volume represents more atherosclerosis. An individual of average health will have a score of 50.
Time Frame: 1 year
Population: all participants with follow up data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Apixaban | Warfarin
Number analyzed (Participants) | 26 | 30
units on a scale | 47 (52) | 54 (120)

ADVERSE EVENTS:
Time Frame: 1 YEAR
Description: same as clinicaltrials.gov
Arm/Group | Apixaban | Warfarin
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes